CLINICAL TRIAL: NCT05596227
Title: Comparison Between Ultrasound Guided Erector Spinae Block vs Thoracolumbar Interfascial Plane Block in Lumbar Spine Surgeries;Randomized Controlled Trial
Brief Title: Ultrasound Guided Erector Spinae Block vs Thoracolumbar Interfascial Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 35634/8/22
Record Dates: First submitted 2022-09-29; First posted 2022-10-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Analgesia; Lumbar Spine Disease
MeSH Terms: conditions — Agnosia; Spinal Diseases | interventions — Propofol; Anesthesia, Intravenous; Fentanyl; Rocuronium; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): Patients will not recieve either erector spinae plane block nor thoracolumbar interfascial plane block
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Rocuronium; Drug: Sevoflurane
- Erector spinae plane block (Active Comparator): Patients will recieve ultrasound guided erector spinae plane block.
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Rocuronium; Drug: Sevoflurane; Other: Erector spinae plane block
- Thoracolumbar interfascial plane block (Active Comparator): Patients will recieve ultrasound guided thoracolumbar interfascial plane block.
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Rocuronium; Drug: Sevoflurane; Other: Thoracolumbar interfascial plane block

INTERVENTIONS:
Drug: Propofol — Induction of anesthesia will be by IV propofol (2-2.5 mg/kg)
  Other Names: Intravenous anesthesia
Drug: Fentanyl — Fentanyl will be injected during the induction of anesthesia (1-1.5 mg/kg)
  Other Names: Intravenous narcotic
Drug: Rocuronium — Rocuronium will be injected during induction of anesthesia (0.6 mg/ kg)
  Other Names: Muscle relaxant
Drug: Sevoflurane — Sevoflurane inhalationa anesthesia will be used for maintainance of anesthesia
  Other Names: Inhalational anesthetic
Other: Erector spinae plane block — In the ESPB group, the probe will be placed in the parasagittal plane at the level of the L3 vertebrae. The spinous process will be visualized, and the probe will move 3 cm laterally from the midline. The erector spinae muscle will be visualized above the transverse process. The needle will be punctured in the craniocaudal direction using the in-plane technique. The needle will be directed superior to the transverse process . Then, 2 mL normal saline solution was injected into the deep fascia of the erector spinae muscle to confirm the proper injection site. After ensuring the location of the needle, 20 mL of 0.25% bupivacaine was administered. The same ESPB procedure will be performed on the other side. In total, 40 mL of 0.25% bupivacaine was administered.
  Arms: Erector spinae plane block
Other: Thoracolumbar interfascial plane block — In the mTLIP group, the probe will be placed vertically at the L3 vertebrae level. The spinous process and the interspinous muscles (i.e., multifidus, longissimus, and iliocostalis) will be visualized as the anatomic guide points. The probe will move laterally to identify the longissimus and iliocostalis muscles. The needle will be inserted between the longissimus and iliocostalis in the medial-to-lateral direction using the in-plane technique. After confirming the location of the needle, 20 mL of 0.25% bupivacaine was administered. The same mTLIP procedure will be performed on the opposite side. In total, 40 mL of 0.25% bupivacaine will be administered.
  Arms: Thoracolumbar interfascial plane block

SUMMARY:
Aim of this Study will be to compare Ultrasound guided erector spinae block vs thoracolumbar interfascial plane (TLIP) block in lumbar spine surgeries.

DETAILED DESCRIPTION:
A total of 180 patients who will be scheduled for single-level lumbar discectomy and laminectomy surgery under general anesthesia will be included in this trial between October 2022 to March 2023.

Inclusion criteria:

The participants will be aged between 20 and 65 years, and will be classified per the American Society of Anesthesiologists (ASA) classification as ASA I-II.

The exclusion criteria Will be a history of coagulation abnormality, anticoagulant treatment, allergies to local anesthetics, skin infections at the site of block area, pregnancy or lactation, and refusal to participate in the study.

A computer program will be used to randomize the participants into 3 groups. Each group (mTLIP block, ESPB, and control) will compose of 60 patients. All patients will be monitored with the standard ASA criteria, electrocardiography, noninvasive blood pressure, and pulse oximetry. Midazolam (2 mg) will be administered intravenously (IV) for sedation. Anesthesia induction will be performed with IV propofol (2-2.5 mg/kg), fentanyl (1-1.5 mg/kg), and rocuronium bromide (0.9 mg/ kg). The patients will be placed in the prone position following intubation. Sevoflurane will be used in a mixture of oxygen and fresh air for anesthesia maintenance. Fentanil will be administered for intraoperative analgesia according to the baseline heart rate and mean arterial pressure of the patients. The intraoperative data (heart rate, peripheral oxygen saturation, noninvasive arterial pressure, and end-tidal carbon dioxide level) will be recorded at 5-minute intervals during the operation. All patients will do lumbar spine surgery by the same surgical team using the same technique.

Block Technique After the induction of anesthesia, either the US-guided mTLIP block or ESPB will be performed in the prone position.A 22G sonovisible block needle with a length of 100 mm will be used to create a puncture. The control group will not receive any intervention. ESPB Technique. In the ESPB group, the probe will be placed in the parasagittal plane at the level of the L3 vertebrae. The spinous process will be visualized, and the probe will move 3 cm laterally from the midline. The erector spinae muscle will be visualized above the transverse process. The needle will be punctured in the craniocaudal direction using the in-plane technique. The needle will be directed superior to the transverse process. Then, 2 mL normal saline solution was injected into the deep fascia of the erector spinae muscle to confirm the proper injection site. After ensuring the location of the needle, 20 mL of 0.25% ropivacaine was administered. The same ESPB procedure will be performed on the other side. In total, 40 mL of 0.25% ropivacaine was administered. mTLIP Technique In the mTLIP group, the probe will be placed vertically at the L3 vertebrae level. The spinous process and the interspinous muscles (i.e., multifidus, longissimus, and iliocostalis) will be visualized as the anatomic guide points. The probe will move laterally to identify the longissimus and iliocostalis muscles. The needle will be inserted between the longissimus and iliocostalis in the medial-to-lateral direction using the in-plane technique. After confirming the location of the needle, 20 mL of 0.25% ropivacaine was administered. The same mTLIP procedure will be performed on the opposite side. In total, 40 mL of 0.25% ropivacaine will be administered. A dose of 1 g paracetamol and 100 mg of tramadol will be administered IV at the end of the surgery to all patients in the mTLIP, ESPB, and control groups. The patients will be extubated after exhibiting sufficient spontaneous respiration and will be transferred to the postanesthesia care unit (PACU). After they attained a modified Aldrete score of 12, the patients will be discharged from the PACU. Standard Postoperative Analgesia Protocol and Measurement of Pain. The postoperative analgesic treatment will be managed using the classic protocol of our department. At the PACU, a fentanyl patient-controlled analgesia (PCA) device will be attached to the patients. The PCA device will be prepared with the following protocol: no infusion dose, a 2-mL (10 µ/ml) bolus, a 20-minute lockout time, and a 4-hour limit of 200 mg. IV 1 g paracetamol was ordered every 6 hours postoperatively. A pain nurse anesthetist, who will be blinded to the trial, will evaluate and record the opioid consumption and the pain scores using a Visual Analog Scale (VAS; 0 = no pain, 10 = the most severe pain). Passive (at rest) and active (while mobilized) VAS scores were recorded at 2, 4, 6, 8 and16 hours during the postoperative period. If VAS was higher than or equal to 4, IV meperidine (0.5 mg/kg) will be administered as rescue analgesia within the postoperative 24-hour period. The opioid-related adverse effects (itching, nausea, vomiting, etc.) and the block procedure times will be also recorded. The block procedure time is defined as the time interval from the start of the visualization of the sonoanatomy to the injection of the local anesthetic solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar spine surgery
* American Society of Anesthesiologists (ASA) classification as ASA I-II.

Exclusion Criteria:

* coagulation abnormality
* anticoagulant treatment,
* allergies to local anesthetics,
* skin infections at the site of block area,
* pregnancy or lactation,
* refusal to participate in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Total postoperative fentanyl requirements | 24 hours
  Total postoperative fentanyl requirements

SECONDARY OUTCOMES:
pain score at rest and during movement | 24 hours
  pain score at rest and during movement using numercal rating score
time of first postoperative analgesic request | 24 hours
  time of first postoperative analgesic request
opioids side effects | 24 hours
  nausea , vomiting, respiratory depression and urine retension

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mohamed Mogahed, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No